CLINICAL TRIAL: NCT04526548
Title: A Multi-center, Prospective Cohort Study on the Diagnostic Value and Prognostic Factors of the RUCAM Scale in Patients With Acute Drug-induced Liver Injury Based on Chronic Liver Disease
Brief Title: A Diagnostic Study on Patients With Drug-induced Liver Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Drug Induced Liver Disease Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: CR2020DILI
Record Dates: First submitted 2020-08-18; First posted 2020-08-26 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Acute Drug-induced Liver Injury; Chronic Liver Disease
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-center, prospective, non-interventional cohort study with an estimated enrollment of 600 patients with acute DILI. According to the inclusion and exclusion criteria, the RUCAM scale and/or expert evaluation, patients with a clinical diagnosis of acute DILI will be included in the study to establish a multi-center, prospective DILI cohort. Depending on the presence or absence of associated chronic liver disease, the patients will be divided into the basic DILI group with chronic liver disease and basic DILI group without chronic liver disease. All enrolled patients should complete at least six months of follow-up.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, non-interventional cohort study with an estimated enrollment of 600 patients with acute DILI. According to the inclusion and exclusion criteria, the RUCAM scale and/or expert evaluation, patients with a clinical diagnosis of acute DILI will be included in the study to establish a multi-center, prospective DILI cohort. Depending on the presence or absence of associated chronic liver disease, the patients will be divided into the basic DILI group with chronic liver disease and basic DILI group without chronic liver disease. All enrolled patients should complete at least six months of follow-up.

This research will propose a new or optimized DILI diagnostic scheme based on the analysis of the problems existing in the practice of RUCAM scale, the clinical characteristics and prognosis of DILI, the exploration of biomarkers, and all the comprehensive information of big data from Hepatox platform, and establish a big data-based diagnosis model or auxiliary diagnosis decision system.

ELIGIBILITY:
Inclusion Criteria:

* No restriction on age and gender.
* Patients need to meet one of the following biochemical thresholds for acute liver injury recommended by the international consensus:

  1. ALT < 5 x ULN
  2. ALP < 2 x ULN
  3. ALT 3 ULN and TBIL 2 ULN
* The duration of liver biochemical abnormalities does not exceed 90 days.
* For the clinical diagnosis of acute drug-induced liver injury, the RUCAM scale ≥ 6 points is required. However, if the RUCAM scale score is 3-5 points, the opinions of 3 experts are needed to confirm the diagnosis of DILI, and the patients can only be enrolled after the experts agree to it.
* The patient signs the informed consent form after fully understanding the nature of the study, the nature of his/her disease, related treatment methods, and the potential risks associated with participating in the trial.

Exclusion Criteria:

* Non-drug induced liver injury
* An inability to complete the visits prescribed by the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with acute drug-induced liver injury
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms and signs | 6 months
  fatigue, anorexia, abdominal distention, jaundice, nausea, vomiting, gingival bleeding, epistaxis, liver pain, hepatomegaly, splenomegaly, fever, rashes, joint pain, skin itching, etc.
Adverse events | 6 months
  Adverse events, severity and time
ALT | 6 months
  U/L
ALP | 6 months
  U/L
TBIL | 6 months
  umol/L